CLINICAL TRIAL: NCT00603837
Title: Thermal Defense of Extremely Low Gestational Age Newborns (ELGANs) During Resuscitation: Exothermic Mattresses vs. Polyethylene Wrap
Brief Title: Warming Mattress Versus Polyethylene Wrapping to Prevent Hypothermia in Preterm Newborns.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Douglas C. Dannaway, Oklahoma University Health Science Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13223
Record Dates: First submitted 2007-12-19; First posted 2008-01-29 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Hypothermia
Keywords: Hypothermia; Prevention; ELGANs(Extremely low gestational age neonates); Polyethylene Wrap; Sodium Acetate Transport Mattress
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blanket (Experimental): This arm includes those Extremely low gestational age newborns (ELGANs) who are to be placed on a sodium acetate warming blanket after delivery.
  Interventions: Device: InfaTherm
- Wrap (Experimental): This arm includes those ELGANs randomized to be wrapped in polyethylene after delivery.
  Interventions: Device: NeoWrap

INTERVENTIONS:
Device: NeoWrap — This is a polyethylene wrap that will be placed around the ELGAN from the neck down to prevent heat loss.
  Arms: Wrap
Device: InfaTherm — A gel blanket containing a sodium acetate-based medium that, when activated, becomes exothermic and provides heat.
  Arms: Blanket

SUMMARY:
Mean axillary temperatures, taken during NICU resuscitation upon admission to the NICU, will not differ between VLBW babies who are occlusively wrapped and very low birth weight (VLBW) babies who are placed on thermal warming blankets.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study will be selected from the inborn population at University Hospital. Eligible patients will be selected from the group of babies with estimated gestational ages of 24-28 weeks and <1250g.

Exclusion Criteria:

* Congenital anomalies with open lesions such as meningomyelocele, or omphaloceles
* Blistering skin conditions
* Resuscitation not performed secondary to infant being below limits of viability as assessed by the in-house attending physician (specifically, according to current NRP recommendations):

  * Where gestation, birth weight, and/or congenital anomalies are associated with almost certain early death, and unacceptably high morbidity is likely among the rare survivors, resuscitation is not indicated. Exceptions may be made based on parental desires.

    * Newborns with confirmed gestation age of less than 24 weeks or birth weight less than 400 grams
    * Anencephaly
    * Confirmed Trisomy 13 or Trisomy 18 syndrome
    * Meconium staining of amniotic fluid
    * Birth assessment of gestational age > 28 weeks or >1250 grams
    * Maternal temp >38 degrees C around the time of delivery.

Ages: 24 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Dannaway, MD, Principal Investigator — University of Oklahoma; Parker L Simon, DO, MPH, Study Director — University of Oklahoma; Marilyn Escobedo, MD, Study Chair — University of Oklahoma
Locations (1):
- Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers were approached on the labor and delivery floor to consent for their child's participation in this study. Recruitment took place from May 2007 to November 2008.
Pre-assignment Details: Three enrolled babies were not included in the analysis. One was found to have a birth weight greater than the cut-off, one was randomized to the wrong group, and one had an unrecorded delivery room temperature.
Groups:
- Blanket: This arm includes those ELGANs who are to be placed on a sodium acetate warming blanket after delivery.
Period: Overall Study
Arm/Group | Blanket | Wrap
Started | 20 | 19
Completed | 17 | 19
Not Completed | 3 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blanket | Wrap | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 19 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39
Temperature [Mean (Standard Deviation); unit: Celsius degrees] | 36.5 (0.67) | 36.1 (0.66) | 36.3 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Intensive Care Unit (NICU) Admission Temperature
Description: Axillary temperature of the infant upon arrival to the neonatal intensive care unit.
Time Frame: At time of admission to the NICU - usually within 10-15 min of birth
Measure: Mean (Standard Deviation); unit: Celsius degrees
Arm/Group | Blanket | Wrap
Number analyzed (Participants) | 17 | 19
Celsius degrees | 36.5 (0.67) | 36.1 (0.66)
Statistical Analysis 1: Comparison: Blanket vs Wrap; Test type: Superiority or Other; p = 0.445, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Blanket | Wrap
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Technical difficulties with the polyethylene wrap were the main limitations (variation of use, heat loss during pulse oximeter adjustment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No